CLINICAL TRIAL: NCT01761812
Title: Determining the Extent and Grade of Prostate Cancer Using MR Elastography, Diffusion Weighted Imaging, and Dynamic Contrast Enhanced MRI With Gadofosveset
Brief Title: Multiparametric MRI for Prostate Cancer Localization and Characterization: New Methods
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate accrual
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Masoom Haider, Staff Radiologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 334-2011
Record Dates: First submitted 2013-01-01; First posted 2013-01-07 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; MRI; Elastography; Gadofosveset
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; gadofosveset trisodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm study (Experimental)
  Interventions: Other: MRI with gadofosveset and MR elastography

INTERVENTIONS:
Other: MRI with gadofosveset and MR elastography

SUMMARY:
The purpose of this study is to determine the ability of several new MRI techniques (MR elastography, dynamic contrast-enhanced MRI with gadofosveset, and oscillating gradient diffusion) to determine the location, size, and grade of prostate carcinoma. Thirty patients with biopsy proven carcinoma awaiting prostatectomy will be included in the study. Ex-vivo MRI will also be conducted on the prostate specimen to obtain high resolution imaging correlates to both in-vivo MRI and whole mount prostatectomy specimens. The investigators hypothesize that the addition of these three techniques will increase the accuracy, sensitivity, and specificity of MRI for detecting clinically significant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* male patients diagnosed with T1C or T2 prostate cancer, awaiting prostatectomy

Exclusion Criteria:

* unable to give informed consent
* contraindication to MRI or MRI contrast agent
* claustrophobia
* renal impairment
* prior hormonal or radiation therapy for prostate cancer
* active prostatitis
* moderate to severe rectal inflammation
* previous rectal surgery
* prostate biopsy within 4 weeks of planned MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient | This outcome measure will be assessed approximately 4 weeks following prostatectomy (an average of 8 weeks from time of enrolment).
  Correlation coefficient between the expected location and grade of prostate cancer as determined by each new MRI method compared with whole mount histological specimen using a 5 mm grid for spatial reference.
Receiver operator characteristic curve for the prediction of prostate cancer for each new MRI method | This outcome measure will be assessed approximately 4 weeks following prostatectomy (an average of 8 weeks from time of enrolment).

CONTACTS AND LOCATIONS:
Overall Officials: Masoom A Haider, M.D., Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada